CLINICAL TRIAL: NCT05069688
Title: Mind the Gaps: Pharmacokinetic Research to Advance Pediatric HIV/TB Cotreatment and TB Prevention
Brief Title: Dolutegravir Pharmacokinetics Among HIV/TB Coinfected Children Receiving Standard and High-dose Rifampicin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: APIN Public Health Initiatives (Unknown); University of Cape Town (Other)
Responsible Party: Principal Investigator, Holly Rawizza, M.D., M.P.H., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002401
Record Dates: First submitted 2021-09-16; First posted 2021-10-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pediatric HIV Infection; Tuberculosis Infection
Keywords: pharmacokinetic; dolutegravir; rifampicin
MeSH Terms: conditions — Latent Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Prospective single-arm, open-label, pharmacokinetic and safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dolutegravir PK during standard and high-dose rifampicin (Experimental): This is a single arm study: all patients are started on HIV/TB cotreatment considered standard of care and then for two weeks (study weeks 20-21) high-dose rifampicin is given during which safety and pharmacokinetics are examined.
  Interventions: Drug: rifampicin

INTERVENTIONS:
Drug: rifampicin — Patients will receive standard TB and HIV treatment, however, for two weeks (study weeks 20-21) the dose of rifampicin will be increased from standard-dose to high-dose to assess pharmacokinetics and safety

SUMMARY:
Tuberculosis (TB) is the leading cause of death among children with HIV, yet insufficient data are available on the pharmacokinetics of newer HIV/TB cotreatment strategies in children. Current WHO-recommended rifampicin dosages result in low concentrations in most children, and high-dose rifampicin may improve outcomes and shorten treatment duration. Yet the impact of high-dose rifampicin on dolutegravir exposures has not been examined in children. This study aims to evaluate the safety and pharmacokinetics of dolutegravir twice daily among HIV/TB coinfected children receiving standard-dose and high-dose rifampicin.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, intensive and sparse pharmacokinetic (PK) and safety study to evaluate steady-state dolutegravir (DTG) concentrations among 20 HIV/TB coinfected children 4 weeks to <6 years of age requiring concurrent TB treatment. Ten patients will be recruited into each of two age cohorts: 4 weeks to <2 years and ≥2 years to <6 years.

Children will be recruited from two large pediatric HIV clinics in Nigeria. Children in this study will receive HIV/TB cotreatment that is considered standard of care consisting of DTG twice daily during rifampicin (RIF)-containing TB treatment. For this portion of the study, the primary intervention is additional blood sampling for drug concentration determination and biomarker assessment. Additionally, during a two week period (study weeks 20-21), the RIF dose will be increased from standard-dose to high-dose RIF, during which two-way PK and toxicity monitoring will occur. Clinical and laboratory monitoring for toxicity during HIV/TB cotreatment is consistent with routine care.

PK sampling for drug concentration determination will occur at three time points during the 48-week study. Specifically, PK sampling will occur at week-20 to evaluate DTG twice daily during standard-dose RIF, week-22 to evaluate DTG twice daily during high-dose RIF, and at week-30 to evaluate DTG once daily after TB treatment is complete.

Additionally, the endogenous biomarker of CYP3A4 activity, 4-beta-hydroxycholesterol to cholesterol ratio, will be evaluated to advance understanding of underlying mechanisms of drug action. Blood sampling to quantify this biomarker will occur at either 4 (among ART-experienced children) or 5 (ART-naive) time points during the 48-week study.

ELIGIBILITY:
Inclusion Criteria:

* ART-naïve or ART-experienced HIV-infected children between 4 weeks and <6 years of age
* Active TB diagnosis
* Weight of at least 3 kilograms
* Consent of the parent or legal guardian

Exclusion Criteria:

* Baseline labs with evidence of ≥grade 3 abnormalities: ALT, total bilirubin, absolute neutrophil count (ANC), platelets, or creatinine
* Suspected TB meningitis or presenting with acute respiratory distress or decompensation
* Receipt of a medication that has drug-drug interactions with dolutegravir or rifampicin

Ages: 4 Weeks to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dolutegravir AUC during standard-dose rifampicin | week 20
  Dolutegravir area under the concentration time curve (AUC) will be compared to therapeutic ranges established in the adult and pediatric literature
Dolutegravir AUC during high-dose rifampicin | week 22
  Dolutegravir AUC will be compared against therapeutic ranges established in the literature and during standard-dose rifampicin

SECONDARY OUTCOMES:
Rifampicin maximum concentration (Cmax) during standard-dose rifampicin | week 20
  Rifampicin Cmax will be determined during standard rifampicin
Rifampicin Cmax during high-dose rifampicin | week 22
  Rifampicin Cmax will be determined during high-dose rifampicin and compared to that observed during standard-dose rifampicin
Proportion of participants experiencing severe (grade 3 or 4) clinical or laboratory adverse events | Week 48
  Laboratory and clinical toxicities are monitored at 8 time points throughout the study and the proportion of children experiencing severe adverse events will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Holly Rawizza, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- University College Hospital/ University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
At the request of researchers de-identified data may be shared.